CLINICAL TRIAL: NCT00959621
Title: Role of LMWH (Enoxaparine) With or Without Aspirin in the Prevention of Habitual Abortion; Special Attention to the Thrombophilic Status of the Mother
Brief Title: Low Molecular Weight Heparin and/or Aspirin in Prevention of Habitual Abortion
Acronym: HABENOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Oulu University Hospital (Other); Karolinska University Hospital (Other); Leiden Hospital, Leiden, The Netherlands (Unknown)
Responsible Party: Professor Risto Kaaja, Helsinki University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HABENOX
Record Dates: First submitted 2009-07-21; First posted 2009-08-14 (Estimated); Last update posted 2009-08-14 (Estimated); Status verified 2009-08

CONDITIONS: Habitual Abortion
Keywords: Habitual abortion; recurrent abortion; hereditary and acquired; thrombophilia; preeclampsia; premature birth; miscarriage; stillbirth; LMWH (low molecular weigh heparin); ASA; aspirin
MeSH Terms: conditions — Abortion, Habitual; Thrombophilia; Pre-Eclampsia; Premature Birth; Abortion, Spontaneous; Stillbirth | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ASA (Active Comparator): The patients received either Enoxaparine+placebo, Enoxaparine+ASA (Aspirin 100 mg) or ASA alone.ASA or placebo were blinded in the two first groups.
  Interventions: Drug: Aspirin
- Klexane (Active Comparator): Clexane (enoxaparine) 40 mg sc
  Interventions: Drug: Klexane
- Aspirin and Enoxaparine (Active Comparator)
  Interventions: Drug: Klexane and ASA

INTERVENTIONS:
Drug: Aspirin — ASA 100 mg once daily per os
  Arms: ASA
Drug: Klexane — Klexane 40 mg sc once daily (HABENOX 1 and 2), Klexane 40 mg twice daily in HABENOX 3
  Arms: Klexane
Drug: Klexane and ASA — Klexane 40 mgx 1 sc and ASA 100 mg po
  Arms: Aspirin and Enoxaparine

SUMMARY:
1 % of all pregnancies end in habitual/recurrent abortion. In about half of women with habitual abortions (HAB) hereditary or acquired (antiphospholipid antibodies) thrombophilia are observed. The investigators wanted to test whether antithrombotic treatment (Low-Molecular Weight Heparin, LMWH, ASA or both combined)would prevent these women from a subsequent abortion. Depending on thrombophilic status the women included in one of the three sub-studies: HABENOX 1 (mild, single thrombophilia), HABENOX 2 (no known thrombophilia), HABENOX 3 (moderate to severe thrombophilia, with combined thrombophilia or moderate to high titer antiphospholipid antibodies).

Study design: Randomised placebo controlled multicenter study.

Number of patients per study: 90 patients per group, 270 altogether.

Timetable: Starting 2/2002, finishing 31.12.2007.

Time frame: >37 weeks of gestation and >24, but <37 weeks of gestation (premature)

Treatment started before 7. gw.

HABENOX 1 and 2:

Study groups:

Group 1 : Enoxaparin 40 mg+ placebo, Group 2: Enoxaparin 40 +ASA 100 mg, Group 3: ASA.

HABENOX 3:

Study groups:

Group 1: Enoxaparin 40 twice daily+ placebo o.d., Group 2: Enoxaparin 40 mg twice daily +ASA 100 mg o.d.

Primary end-points:

Pregnancy outcome: livebirths ( ≥37 weeks of gestation), premature livebirths (≥24, but <37 weeks of gestation)

Secondary end-points: Bleeding complications, intrauterine growth retardation (<-2SD), pre-eclampsia, abruptio placentae,

Ending: In the group of combined medication, tablets will be stopped at 36 weeks of gesta-tion. LMWH will be started in all patients after delivery and continued 6 weeks postpartum.

DETAILED DESCRIPTION:
Background: The prevalence of spontaneous abortions is 1000-1500/10000 pregnancies per year meaning that 10-15% of all pregnancies will end in an abortion; 1/10 of these abortions are recurrent (1 % of all pregnancies). In about half of women with habitual abortions (HAB) hereditary (F V Leiden, F II (prothrombin) mutation, Protein C, S deficiency and anti-thrombin) or acquired (antiphospholipid antibodies) thrombophilia are observed. Efficacy of the medical treatment of patients with a history of HAB has yet to be completely demonstrated. We have recently shown that low-molecular-weight heparin (LMWH) is as effective as unfractionated heparin in prevention of thromboembolic complications in pregnant women and causes less bleeding complications (UFH) and has no osteoporotic effect. LMWH could be safer than UF-heparin during long treatment periods (7-8 months).

Study design: Randomised placebo controlled multicenter study.

Centers: Helsinki (2), Oulu (1), Stockholm (1), Leiden (1)

Number of patients per study: 90 patients per group, 270 altogether

Timetable: Starting 2/2002, finishing 31.12.2007

Drugs:

HABENOX 1 and 2: Study groups Group 1 : Enoxaparin 40 mg+ placebo, Group 2: Enoxaparin 40 +ASA 100 mg, Group 3: ASA.

HABENOX 3: Study groups Group 1: Enoxaparin 40 twice daily+ placebo o.d., Group 2: Enoxaparin 40 mg twice daily +ASA 100 mg o.d.

Time frame: one year since entering the study with primary end-points:livebirths (> 37 weeks of gestation) and premature livebirths (> 24, but <37 weeks of gestation)

Primary end-points: Pregnancy outcome: livebirths (>37 weeks of gestation), premature livebirths (> 24, but <37 weeks of gestation) Secondary end-points: Bleeding complications, intrauterine growth retardation (<-2SD), pre-eclampsia, abruptio placentae,

Inclusion criteria: Three or more consecutive abortions of first trimester (ad h 12+6 wks) or two second trimester abortions (ad h 13 wks-23+6 wks) or one third trimester abortion (24 weeks or more) with one first-second trimester abortions. Depending on the thrombophiliatest (tested before pregnancy) result the patients will included in one of the three sub-studies:

1. HABENOX 1: those who have one thrombophiliatest positive: F V Leiden (heterozygote) or protein C or S deficiency, or anticardiolipin antibodies (low to moderate level), prothrombin gene mutation, or high level of F VIII.
2. HABENOX 2: those with thrombophilia test negative
3. HABENOX 3:those with "high risk" thrombophilia: positive combined thrombophilia, F V Leiden (homozygote), anticardiolipin antibodies (high level >40) , lupusanticoagulant, or AT III deficiency.

During next pregnancy the patient, with inclusion criteria fulfilled, will be asked to sign informed consent and she will be allocated into one of the three treatment groups. The treatment will be started before 7 weeks of gestation. At baseline and follow-up visits plasma, serum and 20 ml morning urine will be frozen (analysed later for antithrombin, protein S, C, APC ratio, PAI1, PAI2, U-PAR, D-dimer, thrombin-antithrombin (TAT) complex, CRP, TNFalpha(+ receptor), ICAM, VEGF(+receptor), urinary stabile metabolites of thromboxane and prostacyclin.

Follow-up: US/Doppler + obstetric check-up at 8, 10, 14, 18, 24, 28, 32 and 36 weeks of gestation Ending: In the group of combined medication, tablets will be stopped at 36 weeks of gesta-tion. LMWH will be started in all patients after delivery and continued 6 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Habenox 1: Three or more consecutive abortions of first trimester (ad h 12+6 wks) or two second trimester abortions (ad h 13 wks-23+6 wks) or one third trimester abortion (24 weeks or more) with one first-second trimester abortions and one thrombophiliatest positive: F V Leiden (heterozygote) or protein C or S deficiency, or anticardiolipin antibodies (low to moderate level), prothrombin gene mutation, or high level of F VIII.
* HABENOX 2: The thrombophilic tests above are negative.
* HABENOX 3:positive combined thrombophilia, F V Leiden (homozygote), anticardiolipin antibodies (high level >40) , lupusanticoagulant, or AT III deficiency.

Exclusion Criteria:

* History of DVT or pulmonary embolism.
* Significant bleeding history.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2002-01; Primary Completion 2004-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pregnancy outcome: livebirths (>37 weeks of gestation), premature livebirths (> 24, but <37 weeks of gestation) | gestational weeks >37 and gestational weeks > 24, but <37

SECONDARY OUTCOMES:
Bleeding complications, intrauterine growth retardation (<-2SD), pre-eclampsia, abruption placenta | gestational weeks > 37 and gestational weeks >24, but <37

CONTACTS AND LOCATIONS:
Overall Officials: Veli-Matti Ulander, MD, Principal Investigator — Helsinki University Hospital, Finland; Laure Morin-Papunen, MD, Study Chair — Oulu University Hospital; Katja Lampinen, MD, Study Chair — Karolinska University Hospital; Kitty Bloemenkamp, MD, Study Chair — Leiden University Hospital, Leiden, The Netherlands; Janvier Visser, MD, Study Chair — Leiden University Hospital, Leiden, The Netherlands
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Hamulyak EN, Scheres LJ, Marijnen MC, Goddijn M, Middeldorp S. Aspirin or heparin or both for improving pregnancy outcomes in women with persistent antiphospholipid antibodies and recurrent pregnancy loss. Cochrane Database Syst Rev. 2020 May 2;5(5):CD012852. doi: 10.1002/14651858.CD012852.pub2. PMID 32358837